CLINICAL TRIAL: NCT04112719
Title: Assessing Effects of Lateral Tilt on Cardiac Output Using a Non-invasive Technique
Acronym: LATCOIN
Status: Completed | Type: Observational
Sponsor: The University of Texas Medical Branch, Galveston (Other)
Responsible Party: Sponsor
Other Study IDs: 19-0086
Record Dates: First submitted 2019-09-24; First posted 2019-10-02 (Actual); Last update posted 2020-10-26 (Actual); Status verified 2019-09

CONDITIONS: Cardiac Output
MeSH Terms: interventions — Supine Position

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Control arm/pregnant patients at term: Control arm where the term pregnant patient will be lying on the bed at 45 degrees.
- Experimental/Supine: Term pregnant patient will be positioned in supine. Changes in hemodynamics will be measured.
  Interventions: Other: supine position
- Experimental/15 degrees lateral tilt: Term pregnant patient will be positioned at 15 degrees in lateral tilt. Changes in hemodynamics will be measured.
  Interventions: Other: 15 degrees lateral tilt
- Experimental/30 degrees lateral tilt: Term pregnant patient will be positioned at 30 degrees in lateral tilt. Changes in hemodynamics will be measured.
  Interventions: Other: 30 degrees lateral tilt

INTERVENTIONS:
Other: supine position — The patient will be placed in a supine position. Changes in cardiac output will be measured.
  Groups: Experimental/Supine
Other: 15 degrees lateral tilt — The patient will be placed in 15 degrees lateral tilt position. Changes in cardiac output will be measured.
  Groups: Experimental/15 degrees lateral tilt
Other: 30 degrees lateral tilt — The patient will be placed in 30 degrees lateral tilt position. Changes in cardiac output will be measured.
  Groups: Experimental/30 degrees lateral tilt

SUMMARY:
In pregnant term patients, we intent to use a non invasive cardiac output monitor to detect the changes in cardiac output as the patient is being placed in different positions.

The patient will be placed on her back, flat, and in left lateral tilt at two different angles. Measurements of cardiac output will be recorded.

DETAILED DESCRIPTION:
Aortocaval compression compromising tissue perfusion has always been of a concern in term pregnant women undergoing caesarian delivery or regional anesthesia when placed in the supine position. It is believed that this phenomena happens when the gravid uterus compresses the inferior vena cava (IVC)resulting in decreased venous return and hence cardiac output (CO) leading to low placental perfusion and associated fetal heart rate changes.

Hence, due to these concerns, left lateral tilt is currently a common practice in obstetrics and it is believed to relief aortocaval compression and to improve blood flow to the fetus.

Supporting evidence for this intervention remains controversial, and shows conflicting results. Some studies suggest that lateral tilt does not affect neonatal outcomes (1) or changes in cardiac output in patients with no regional anesthesia (2). While others suggest it can actually increase the volume of the IVC, especially when the patient is tilted 30 degrees or more (3) and may lead to increases in CO (4).

Non-invasive hemodynamic monitoring (NICOM, Cheetah Medical), an FDA approved device, is currently being used to detect changes in CO in the United States. Its use has been validated in different clinical settings (5,6).

Our hypothesis is that CO is increased in pregnant women that were placed in the lateral tilt position.

We intend to compare CO measurements using the non-invasive hemodynamic monitoring among term pregnant patients in supine vs lateral tilt position.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women between the ages of 18-50.
* Elective repeat cesarean section or induction of labor.

Exclusion Criteria:

* Incarcerated patients
* Patient unwilling or unable to provide consent
* Intrauterine fetal demise (no fetal heart beat identified and documented by two physicians).

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Pregnant women
Study Population: Term Pregnant women presenting for delivery
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2019-11-01 (Actual); Primary Completion 2020-04-01 (Actual); Study Completion 2020-04-01 (Actual)

PRIMARY OUTCOMES:
Cardiac output (liters/minute) | 20 minutes
  Changes in cardiac output while lying on bed at 45 degrees
Cardiac output (liters/minute) | 20 minutes
  Changes in cardiac output while patient in placed in supine position
Cardiac output (liters/minute) | 20 minutes
  Changes in cardiac output while patient in placed in lateral tilt at 15 degrees
Cardiac output (liters/minute) | 20 minutes
  Changes in cardiac output while patient in placed in lateral tilt at 30 degrees

SECONDARY OUTCOMES:
Blood pressure (mm Hg) | 80 minutes
  Changes in blood pressure while patient in placed in different positions
Fetal heart rate abnormalities (beats/minute) | 80 minutes
  Changes in fetal heart rate tracing while patient is placed in different positions

CONTACTS AND LOCATIONS:
Overall Officials: Antonio Saad, MD, Study Director — UTMB
Locations (1):
- UTMB, Galveston, Texas, United States

IPD SHARING:
Plan to Share IPD: No